CLINICAL TRIAL: NCT06338566
Title: Prospective Follow-up of Functional, Bone and Septic Results of Ankle Arthrodesis With Transplanted Nail
Brief Title: Prospective Follow-up of the Results of Nail Arthrodesis of the Ankle
Acronym: PROCLOU
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PPRC10; 2023-A01975-40 (Other: IDRCB)
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up — Follow-up at D45, 3 months and 6 months, with scoring, radiological monitoring and assessment of wound healing

SUMMARY:
The goal of this prospective, single-center observational study is to describe the functional outcome of the surgical procedure in patient who undergone transplanted centromedullary nailing in the septic setting.

Patients will be asked to complete a questionnaire during follow-up consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years
* having undergone septic nailing in the operating theatre
* with social security coverage

Exclusion Criteria:

* Patient with 6-month follow-up not possible (medical wandering, transient patient),
* Patient who has benefited from another means of osteosynthesis
* Patients whose long-term return to weight-bearing will not be possible for reasons other than ankle arthrodesis surgery.
* Persons able to give consent but unable to read or write French
* Opposes participation in the study
* Patients whose cognitive capacity does not allow them to answer questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent ankle surgery and have an ankle arthrodesis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
bony outcome of transcalcaneal nailing | up to 6 months
  percentage of patients with aseptic consolidation at 6 months post-op

SECONDARY OUTCOMES:
functional result of the procedure | up to 6 months
  percentage of patients able to walk again at 6 months post-op

IPD SHARING:
Plan to Share IPD: No